CLINICAL TRIAL: NCT05960292
Title: Laparoscopic Versus Vaginal Approach Closure Complications of Vaginal Vault in Laparoscopic Hysterectomy
Brief Title: Laparoscopic Versus Vaginal Approach Closure Complications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mohamed Adel Hussien
Record Dates: First submitted 2023-07-12; First posted 2023-07-25 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Vaginal Vault Prolapse
Keywords: Laparoscopic hysterectomy; Vaginal hysterectomy
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Laparoscopy; Hysterectomy, Vaginal

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaginal Hysterectomy (Group) (Active Comparator): About 28 female patients will have vaginal vault closure by vaginal approach
  Interventions: Procedure: Laparoscopic and Vaginal Hysterectomy
- Abdominal Laparoscopic Hysterectomy (Group) (Active Comparator): About 28 female patients will have vaginal vault closure by Abdominal Laparoscopic approach
  Interventions: Procedure: Laparoscopic and Vaginal Hysterectomy

INTERVENTIONS:
Procedure: Laparoscopic and Vaginal Hysterectomy — To make a comparison between the Vaginal Vault complications after Hysterectomy

SUMMARY:
Hysterectomy is considered as a common operation in Gynecology. Hysterectomy could be made by vaginally, laparoscopically or abdominally. The American Congress of Obstetricians and Gynecologist advises the use of a minimally invasive technique for the sake of women and to decrease hospital stay and costs.

DETAILED DESCRIPTION:
Laparoscopic hysterectomy (LH) is a minimally invasive operation that could be made when vaginal hysterectomy is not accessible due to anatomical problems.

Vaginal cuff dehiscence (VCD) is a severe adverse event and occurs more frequently after total laparoscopic hysterectomy (TLH) compared with abdominal and vaginal hysterectomy.

The study shows effects of the laparoscopic approach versus the vaginal route for the management of vaginal cuff closure during total laparoscopic hysterectomy on female sexual function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who undergo laparoscopic hysterectomy
2. Age ranged from 40 to 80 years.
3. Patients suffering from chronic pelvic inflammatory disease (PID)
4. Dysfunctional uterine bleeding
5. Adenomyosis
6. Endometriosis
7. Fibroid
8. Endometrial hyperplasia
9. Benign ovarian cyst

Exclusion Criteria:

* Patients with known malignancy

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Post operative bleeding (defined as blood loss ≥500 cc) | First 24 hours after The Operations
  Amount of lost blood will be measured in terms of assessment of Hemoglobin and Hematocrit levels before and after operation.
Postoperative pain | First 24 hours after The Operations
  Assessment of the pain post-operatively in patients with pain score as : Total scores vary from 0 to 10 in this method, with a higher score indicating more severe pain

CONTACTS AND LOCATIONS:
Overall Officials: ElSayed ElDesouky, Assist.Prof., Principal Investigator — Al-Azhar University, Faculty of medicine for boys
Locations (1):
- Al-Azhar University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided